CLINICAL TRIAL: NCT00491465
Title: Randomized,Controlled,Open,Cross-Over Intervention Study for Evaluating the Role of Physical Activity in the Treatment of Children With Type 1 Diabetes.
Brief Title: The Role of Physical Activity in the Treatment of Children With Type 1 Diabetes.
Acronym: 4301
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: rmc074301ctil
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes, physical activity, pediatric, metabolic control
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Intensive Physical activity
Behavioral: Control- regular physical activity

SUMMARY:
Randomized, controlled, open, comparative intervention study in two groups, each consisting of 25 children with type 1 diabetes that will undergo twelve weeks of exercise program (intensive arm) and twelve weeks of regular activity (non intensive arm) separated by four week of washout period. The study will be conducted in a crossover manner: one group starting with the intensive arm followed by the non intensive arm and vice versa. Blood glucose, HbA1C, Fructosamine, 3 days continuous glucose monitoring system (CGMS), total daily insulin dose, fasting lipid profile, body impedance and BMR will be measured. Self esteem and quality of life questionnaires will be filled.

DETAILED DESCRIPTION:
Randomized, controlled, open, comparative, cross-over, intervention study in 50 children with type 1 diabetes.

objectives:

Primary objective To evaluate the efficacy and safety of physical activity for metabolic control in children with type I diabetes.

Secondary objectives

1. To characterize the severity and pattern of occurrence of hypo and hyperglycemic episodes during and after exercise program in type I diabetic children.
2. To evaluate changes in insulin sensitivity during and after periods of exercise in type I diabetic children.
3. To evaluate the short term effect of exercise on BMI and body composition in type I diabetic children.
4. To evaluate the short term effect of exercise on lipid profile in type I diabetic children.
5. To evaluate differences in self esteem and quality of life between exercising and non exercising type I diabetic children.

Randomization:

Children will be randomly allocated into two groups of 25.The study will be conducted in a crossover manner:one group starting with the intensive arm followed by the non intensive arm and vice versa.

methods:

1. The study will have an intensive arm and a non intensive arm, each lasting 12 weeks.
2. Children fulfilling the inclusion and exclusion criteria will be randomly assigned to two groups. Each group will include 25 patients.
3. Participants will fill questionnaires regarding physical activity.
4. The first group will start with the intensive arm, followed by one month washout, and then the non intensive arm.
5. The second group will start the study with the non intensive arm, followed by one month washout and then the intensive arm .
6. The intensive arm will consist of an exercise program which will include high intensity progressive exercise (75% maximum age adjusted heart rate HRmax) 3 days a week for 90 minutes. The 90 min exercise will be a combination of aerobic exercise 45min. and resistance exercise 45 min.
7. The exercise program will be planned and carried out by professional sports instructors.
8. During the non intensive arm the participants will resume regular daily activity. They will keep records of their weekly physical activity and will get a weekly phone call from the treating doctor, addressing specifically physical activity performed during the past week and glucose levels before and after exercise.
9. The following parameters will be measured for both groups at the beginning and the end of the intensive and non intensive arm and once again 12 weeks afterwards : Weight, height, pulse, blood pressure, waist circumference, skin folds, HbA1C , fructosamine ,3 days CGMS +3 day SBGM profile (will be measured to 40% of participants chosen randomly) ,total daily insulin dose ,blood sample for fasting lipid profile ,Body impedance and BMR , self esteem and quality of life questionnaires .
10. Study participants will be required to measure blood glucose by glucometer at least 4 times a day and to record hypo and hyperglycemic events and their severity.

15.Both children and investigators will be blinded to CGMS results. 16.During the 3 day CGMS recording, the children's parents will be asked to monitor SBGM once during the night (in the intensive arm, following the exercise day).

ELIGIBILITY:
Inclusion Criteria:

1. Type I diabetic children
2. Tanner stage II-IV
3. Patients of the Schneider's national institute of childhood diabetes. Duration of diabetes
4. more than one year.
5. HbA1C between 8 and 12 at time 0.
6. Mandatory 4 daily self blood glucose measurements and daily recording of adverse events.
7. A signed informed consent of the parents and child.

Exclusion Criteria:

1. Additional chronic significant disease such as cardiac, liver, renal disease .
2. Children who exercise regularly more than 180 min per week.
3. Cardiac symptoms: history of chest pain , syncope , palpitations or dyspnea during exercise.
4. Eating disorders.
5. Participation in a study during the past month.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2007 (Estimated)
Dates: Start 2007-07; Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
HbA1C | 0,3 monthes
fructosamine | 0,3 monthes

SECONDARY OUTCOMES:
Body composition & BMR | 0,3 monthes
Self esteem & QOL questionnaires | o, 3 monthes
3 days CGMS & SBGM profile | 0,3 monthes

CONTACTS AND LOCATIONS:
Overall Officials: Ravital Nimri, MD, Principal Investigator — Rabin Medical Center; Moshe Phillip, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Schnider children's medical center, Petah Tikva, Israel